CLINICAL TRIAL: NCT01068028
Title: Safety, Tolerability and Pharmacokinetics of Multiple Escalating Doses of ORM-12741
Brief Title: Safety and Pharmacokinetic Study With Multiple Ascending Doses of ORM-12741
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Jutta Hänninen / Clinical Study Manager, Orion Corporation, Orion Pharma
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3098008
Record Dates: First submitted 2010-02-10; First posted 2010-02-12 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Healthy volunteer study
MeSH Terms: interventions — ORM-12741

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo for ORM-12741 (Placebo Comparator)
  Interventions: Drug: Placebo for ORM-12741
- ORM-12741 (Experimental)
  Interventions: Drug: ORM-12741

INTERVENTIONS:
Drug: ORM-12741 — Ascending multiple doses to sequential panels
  Arms: ORM-12741
Drug: Placebo for ORM-12741
  Arms: Placebo for ORM-12741

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of multiple ascending doses of ORM-12741.

DETAILED DESCRIPTION:
The purpose is to evaluate the safety, tolerability and pharmacokinetics of escalating multiple doses of ORM-12741 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Good general health ascertained by detailed medical history and physical examinations.
* Males between 18 and 45 years (inclusive).
* Body mass index (BMI) between 18-30 kg/m2 inclusive (BMI = weight/height2).
* Weight 55-100 kg (inclusive).

Exclusion Criteria:

* Evidence of clinically significant cardiovascular, renal, hepatic, haematological, gastro-intestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric disease as judged by the investigator.
* Any condition requiring regular concomitant medication including herbal products or likely to need any concomitant medication during the study.
* Susceptibility to severe allergic reactions.
* Regular consumption of more than 14 units of alcohol per week (1 unit = 4 cl spirits, about 13 g of alcohol).
* Current use of nicotine-containing products more than 5 cigarettes or equivalent/day.
* Inability to refrain from using nicotine-containing products during the stay at the study centre.
* Inability to refrain from consuming caffeine-containing beverages during the stay at the study centre e.g. propensity in getting headache when refraining from caffeine-containing beverages.
* Blood donation or loss of significant amount of blood within 3 months prior to the screening visit.
* Abnormal finding in ECG, vital signs, laboratory tests or physical examination.
* Intake of an investigational compound within 3 months prior to the start of this study or earlier participation in a clinical study with ORM-12741

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety measures, i.e. assessing adverse events, vital signs, ECG, safety laboratory values | 12 days

SECONDARY OUTCOMES:
Pharmacokinetic profile (Cmax, tmax, t1/2, AUC, PTF) of ORM-12741 and its metabolites | PK samples will be collected for 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Déborah Metzger, MD, Principal Investigator — Forenap Pharma
Locations (1):
- Forenap Pharma, Rouffach, France